CLINICAL TRIAL: NCT05358977
Title: Fibrin Sealant to Reduce Postoperative Bleeding After Blepharoplasty
Brief Title: Fibrin Sealant in Eyelid Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB21-0341
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Blepharoptosis; Ecchymosis; Eyelid
MeSH Terms: conditions — Blepharoptosis; Ecchymosis | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Intervention Model Description: Each participant in the study will receive a topical application of fibrin sealant (Tisseel) in one of their upper eyelid eyelid blepharoplasty closures in addition to standard blepharoplasty closure techniques. The other eyelid will receive standard blepharoplasty closure techniques alone, without fibrin sealant. Both sides will receive 1 minute of pressure, after application of Tisseel, to mask which side received treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: At the end of the intervention, both sides will receive 1 minute of pressure to mask the patient as to which side received treatment. Postoperative photographs will be assessed by two masked ophthalmic surgeons who will rate the degree of postoperative bruising. Upper and lower eyelids of each patient will be evaluated separately. Observers will assess each side for ecchymosis using a 10-point Likert scale (1, none; 10, severe) on postoperative days 1, 3 and 7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tisseel (Experimental): Patients are undergoing bilateral blepharoplasty. In this arm (Tisseel), the patient with undergo blepharoplasty with topical Tisseel placed in the incision prior to standard closure. 1 minute of pressure will be exerted to both eyelids after closure to mask the patient as to which eyelid received the Tisseel.
  Interventions: Biological: Tisseel
- Control (No Intervention): Patients are undergoing bilateral blepharoplasty. In this arm (Control), the patient with undergo blepharoplasty with standard closure along. 1 minute of pressure will be exerted to both eyelids after closure to mask the patient as to which eyelid received the Tisseel.

INTERVENTIONS:
Biological: Tisseel — Intraoperatively, the intervention side will receive topical administration of Tisseel to the blepharoplasty incision. A 2mL syringe of Tisseel product will be used as per the product monograph for an area of < 8cm2. There will be no variation in surgical counselling or technique, with the exception of the use of Tisseel in one eyelid closure. Both eyelids will otherwise receive standard blepharoplasty surgical techniques. There will be no monitoring of compliance necessary, given the Tisseel will be utilized intraoperatively.
  Arms: Tisseel

SUMMARY:
This study is looking at the effect of Tisseel in eyelid surgery. Fibrin sealants (Tisseel) cause there to be less bleeding during surgery. Surgeons have used Tisseel for over two decades to reduce bruising. Ophthalmologists use it during surgery. Yet, there are no studies confirming the effect of Tisseel during eyelid surgery. Unpublished work suggests that it is effective in decreasing postoperative bruising. This study will confirm the effect of Tisseel on postoperative bruising in blepharoplasty.

DETAILED DESCRIPTION:
The study is designed as a superiority randomized control trial. Tisseel will be used for hemostasis during the closure of one blepharoplasty incision. The side to receive Tisseel will be determined using a random number generator. After application of topical Tisseel, both eyelids will undergo standard blepharoplasty closure techniques. Pressure will be placed on both upper eyelids to mask the patient as to what side received the Tisseel.

Postoperatively, patients will take photographs on postoperative days 1, 3, 7. Photographs with poor quality not allowing accurate assessment will not be scored and that visit will not be included in the study. The photographs will be assessed by two masked ophthalmic surgeons who will rate the degree of postoperative bruising. Upper and lower eyelids of each patient will be evaluated separately. Observers will assess each side for ecchymosis using a 10-point Likert scale (1, none; 10, severe) on postoperative days 1, 3 and 7.

Given a blepharoplasty costs the healthcare system approximately $950 Canadian dollars, a vial of Tisseel ($160) would add approximately 17% to the cost (160/942.43 = 16.97%). Therefore, a 17% percent margin of superiority was used in power calculations to determine statistical efficacy of the intervention.

A power calculation for a randomized control superiority trial was performed. A 17% percent margin of superiority was used in power calculations. These variable were used to calculate for a dichotomous outcome superiority trial. The calculated sample size was calculated to be 27 in each group.

Tisseel is made from human plasma and may therefore contain infectious agents, such as viruses, that can cause disease. With over two decades of use, there has never been a reported case of hepatitis (HAV, HBV, HCV) or human immunodeficiency virus (HIV) transmission. However, Tisseel used during thoracic surgery has been associated with increased seropositivity for parvovirus B19. Although there were no complications associations with the parvovirus B19 infection observed, infection with parvo B19 can theoretically cause anemia or arthralgias, fifth disease in children, miscarriage, or rash. All patients who would be at risk of complications from such an infection were excluded.

Research is ongoing, despite the continuation of the COVID-19 pandemic. Postoperative photographs taken by the patients are used to minimize contact during care.

ELIGIBILITY:
Inclusion Criteria:

• Patient undergoing bilateral upper eyelid blepharoplasty

Exclusion Criteria:

* Hypersensitivity to the fibrin adhesive or components of it
* Religious belief prohibiting the use of blood products
* Pregnancy
* Immunodeficiency
* Age ≤18 years of age
* Breastfeeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Bruising as defined by masked observers using a 10-point Likert scale. | 1 week
  Postoperative photographs will be assessed by two masked ophthalmic surgeons who will rate the degree of postoperative bruising. Upper and lower eyelids of each patient will be evaluated separately. Observers will assess each side for ecchymosis using a 10-point Likert scale (1, none; 10, severe) on postoperative days 1, 3 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Punja, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson DF, Letassy NA, Thompson GD. Fibrin glue: a review of its preparation, efficacy, and adverse effects as a topical hemostat. Drug Intell Clin Pharm. 1988 Dec;22(12):946-52. doi: 10.1177/106002808802201203. PMID 2468466
- [Background] Sowerby L, Kim LM, Chow W, Moore C. Intra-operative nasal compression after lateral osteotomy to minimize post-operative Peri-orbital ecchymosis and edema. J Otolaryngol Head Neck Surg. 2019 Oct 16;48(1):50. doi: 10.1186/s40463-019-0370-7. PMID 31619274
- [Background] Zoumalan R, Rizk SS. Hematoma rates in drainless deep-plane face-lift surgery with and without the use of fibrin glue. Arch Facial Plast Surg. 2008 Mar-Apr;10(2):103-7. doi: 10.1001/archfaci.10.2.103. PMID 18347237
- [Background] Marchac D, Greensmith AL. Early postoperative efficacy of fibrin glue in face lifts: a prospective randomized trial. Plast Reconstr Surg. 2005 Mar;115(3):911-6; discussion 917-8. doi: 10.1097/01.prs.0000153219.32665.d5. PMID 15731694
- [Background] Panda A, Kumar S, Kumar A, Bansal R, Bhartiya S. Fibrin glue in ophthalmology. Indian J Ophthalmol. 2009 Sep-Oct;57(5):371-9. doi: 10.4103/0301-4738.55079. PMID 19700876
- [Background] Horowitz B, Busch M. Estimating the pathogen safety of manufactured human plasma products: application to fibrin sealants and to thrombin. Transfusion. 2008 Aug;48(8):1739-53. doi: 10.1111/j.1537-2995.2008.01717.x. Epub 2008 May 7. PMID 18466171
- [Background] Kawamura M, Sawafuji M, Watanabe M, Horinouchi H, Kobayashi K. Frequency of transmission of human parvovirus B19 infection by fibrin sealant used during thoracic surgery. Ann Thorac Surg. 2002 Apr;73(4):1098-100. doi: 10.1016/s0003-4975(02)03415-x. PMID 11996248